CLINICAL TRIAL: NCT02307656
Title: Assessment of the Taste Properties of Atazanavir and Cobicistat and Pediatric Oral Test Formulations Containing Both Atazanavir and Cobicistat in Healthy Adults
Brief Title: Taste Properties of Atazanavir and Cobicistat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AI424-517
Record Dates: First submitted 2014-10-29; First posted 2014-12-04 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: HIV in Adults
MeSH Terms: interventions — Atazanavir Sulfate; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atazanavir and Cobicistat (Other): Stage 1:Taste evaluation using Active Pharmaceutical Ingredient (API)
  Stage 2:Taste Optimization using API (flavours and sweeteners)
  Stage 3:Prototypes of the API - containing clinical trial materials
  Interventions: Drug: Atazanavir; Drug: Cobicistat; Drug: Active Pharmaceutical Ingredient

INTERVENTIONS:
Drug: Atazanavir
Drug: Cobicistat
Drug: Active Pharmaceutical Ingredient
  Other Names: (API)

SUMMARY:
The primary objective is to assess the taste properties of atazanavir (ATV) and cobicistat (COBI) alone and in combination as well as oral test formulations containing both ATV and COBI.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men and women, ages ≥18 years
* Subjects who are qualified professional sensory panelists
* Healthy subjects as determined by no clinically significant deviation from normal in medical history and physical assessment

Exclusion Criteria:

* Any acute or chronic condition that may alter taste or smell sensory perception
* Any significant acute or chronic medical illness or any surgery within 4 weeks of the study drug administration
* Positive HIV test using an oral swab kit (such as OraQuick®) to detect HIV-1 or -2 antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Taste properties of ATV & COBI alone & in combination as well as oral test formulations containing both ATV & COBI Aromatic identity will be measured using the Flavor Profile of the Flavor Leadership Criteria | Every 6 weeks from the time of subject enrollment up to 2 years
Taste properties of ATV & COBI alone & in combination as well as oral test formulations containing both ATV & COBI amplitude will be measured using the Flavor Profile of the Flavor Leadership Criteria | Every 6 weeks from the time of subject enrollment up to 2 years
Taste properties of ATV & COBI alone & in combination as well as oral test formulations containing both ATV & COBI mouth-feel will be measured using the Flavor Profile of the Flavor Leadership Criteria | Every 6 weeks from the time of subject enrollment up to 2 years
Taste properties of ATV & COBI alone & in combination as well as oral test formulations containing both ATV & COBI off-notes will be measured using the Flavor Profile of the Flavor Leadership Criteria | Every 6 weeks from the time of subject enrollment up to 2 years
Taste properties of ATV & COBI alone & in combination as well as oral test formulations containing both ATV & COBI aftertaste will be measured using the Flavor Profile of the Flavor Leadership Criteria | Every 6 weeks from the time of subject enrollment up to 2 years

OTHER OUTCOMES:
Incident of adverse events will be tabulated and reviewed for potential significance and clinical important | Approximately up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Senopsys Llc, Woburn, Massachusetts, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm